CLINICAL TRIAL: NCT06478693
Title: A Phase 1, Open-Label, First-in-Human, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of MT-303 in Adults With Advanced or Metastatic GPC3-Expressing Cancers, Including Hepatocellular Carcinoma
Brief Title: A Study of MT-303 in Adults With Advanced or Metastatic GPC3-Expressing Cancers, Including HCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Myeloid Therapeutics (Industry)
Collaborators: CREATE Medicines (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MTX-GPC3-303
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver Cancer; Hepatocellular Carcinoma (HCC); Glypican-3; Chimeric antigen receptor; CAR-M
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Simpson-Golabi-Behmel syndrome | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT-303 (Experimental): Participants will receive MT-303 through intravenous infusion.
  Interventions: Drug: MT-303
- MT-303 + Atezolizumab + Bevacizumab (Experimental): Participants will receive MT-303 in combination with Atezo/Bev through intravenous infusion.
  Interventions: Drug: MT-303 +Atezolizumab + Bevacizumab

INTERVENTIONS:
Drug: MT-303 — MT-303
  Arms: MT-303
Drug: MT-303 +Atezolizumab + Bevacizumab — MT-303 in combination with Atezo/Bev
  Arms: MT-303 + Atezolizumab + Bevacizumab

SUMMARY:
This is a multicenter, open-label, Phase 1, first-in-human, dose-escalation study designed to assess the safety, tolerability and define the RP2D of MT-303 alone (Module 1) and in combination with Atezo/Bev (Module 2) in participants with advanced hepatocellular carcinoma expressing GPC3.

DETAILED DESCRIPTION:
Participants will be enrolled into one of two treatment modules:

* Module 1 (Monotherapy): Participants will receive MT-303.
* Module 2 (Combination therapy): Participants will receive MT-303 in combination with atezolizumab + bevacizumab (Atezo/Bev).

In Module 1 (Monotherapy), participants will receive MT-303 across five dose-escalation cohorts and in Module 2 (Combination therapy), participants will receive MT-303 in combination with Atezo/Bev across five dose-escalation cohorts.

Additional cohorts in both modules may be scheduled based on emerging safety and PK data.

Participants will be sequentially enrolled into Cohorts 1 through 5. Both modules will be enrolled concurrently, with Module 2 dosing beginning at one dose level below the known safe dose in Module 1. Safety Review Committee decisions will be informed by all available safety data from Modules 1 and 2.

ELIGIBILITY:
Inclusion Criteria

* Aged 18 years or older
* Histological diagnosis of advanced/recurrent or metastatic and/or unresectable HCC. [Note: participants with other tumor types expressing GPC3 may be eligible for Module 1 pending a discussion with the Medical Monitor. Only participants with HCC are eligible for Module 2.
* Measurable lesion per RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Child-Pugh score: Class A
* Adequate organ function

General Exclusion Criteria

* Known active CNS metastasis and/or carcinomatous meningitis.
* Any acute illness including active infection
* History of liver transplantation or on waiting list
* Participants with untreated or incompletely treated varices with bleeding or high risk for bleeding
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* History of symptomatic congestive heart failure
* History of chronic or recurrent (within the last year) severe autoimmune or immune mediated disease requiring steroids or other immune-suppressive treatments.

Additional Module 2 Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Significant cardiovascular disease
* History of severe hypersensitivity to atezolizumab and/or bevacizumab.
* History of idiopathic pulmonary fibrosis
* Prior history of hypertensive crisis or hypertensive encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Type, incidence and severity of Adverse Events | Up to 2 years from the last dose of Investigational Medicinal Product (IMP)
  Safety and tolerability profile assessed by the Common Terminology Criteria for Adverse Events v5.0
Recommended Phase 2 Dose (RP2D) | 28 days from the last dose of IMP
  The RP2D will be determined using dose limiting toxicities (DLTs) and all other available study data
Optimal Biological dose (OBD) | 21 days from the last dose of IMP
  The OBD will be determined using dose limiting toxicities (DLTs) and all other available study data
Change from baseline in vital signs | Up to 30 days from the last dose of IMP
  Temperature, weight, height, pulse rate and blood pressure will be assessed
Change in laboratory parameters | Up to 30 days from the last dose of IMP
  Hematology, chemistry, coagulation, virology and urine analysis will be assessed.
Change from baseline in ECG parameters | Screening, Day 1 and Day 15

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Day 1, 2, 3, 8, 15 and once every 28 days post first dose of IMP for Module 1 and Day 1, 2, 8 and once every 21 days post first dose of IMP for Module 2.
  PK parameter: Plasma concentrations
Pharmacokinetics (PK) | Day 1, 2, 3, 8, 15 and once every 28 days post first dose of IMP for Module 1 and Day 1, 2, 8 and once every 21 days post first dose of IMP for Module 2.
  PK parameter: Area under Curve
Pharmacokinetics (PK) | Day 1, 2, 3, 8, 15 and once every 28 days post first dose of IMP for Module 1 and Day 1, 2, 8 and once every 21 days post first dose of IMP for Module 2.
  PK parameter: Time of maximum observed plasma concentration (tmax)
Pharmacokinetics (PK) | Day 1, 2, 3, 8, 15 and once every 28 days post first dose of IMP for Module 1 and Day 1, 2, 8 and once every 21 days post first dose of IMP for Module 2.
  PK parameter: Plasma Clearance (CL)
Pharmacokinetics (PK) | Day 1, 2, 3, 8, 15 and once every 28 days post first dose of IMP for Module 1 and Day 1, 2, 8 and once every 21 days post first dose of IMP for Module 2.
  PK parameter: Volume of Distribution (Vd)
Pharmacokinetics (PK) | Day 1, 2, 3, 8, 15 and once every 28 days post first dose of IMP for Module 1 and Day 1, 2, 8 and once every 21 days post first dose of IMP for Module 2.
  PK parameter: Mean residence time (MRT)
Pharmacokinetics (PK) | Day 1, 2, 3, 8, 15 and once every 28 days post first dose of IMP for Module 1 and Day 1, 2, 8 and once every 21 days post first dose of IMP for Module 2.
  PK parameter: terminal rate constant (λz)
To assess adverse events of special interest (AESI) by measuring infusion reaction | upto 2 years from the last dose of IMP
To assess adverse events of special interest (AESI) by measuring cytokine release syndrome (CRS) | Up to 2 years from the last dose of IMP
To assess adverse events of special interest (AESI) by measuring immune effector cell-associated neurotoxicity syndrome (ICANS) | Up to 2 years from the last dose of IMP
To assess adverse events of special interest (AESI) by measuring hypersensitivity reaction | Up to 2 years from the last dose of IMP
To assess adverse events of special interest (AESI) by checking for second primary malignancy | upto 2 years from the last dose of IMP

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Maurer, MD, Study Director — Myeloid Therapeutics
Locations (9):
- Australia (4):
  - St Vincent's Hospital, Sydney, New South Wales
  - Integrated Clinical Oncology Network (ICON) Pty Ltd, Woolloongabba, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Murdoch, Western Australia
- South Korea (3):
  - Pusan National Univesity Hospital, Busan
  - Cha University Bundang Medical Center, Gyeonggi-do
  - Seoul National University Hospital, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Tzu Chi Hospital, Taipei